CLINICAL TRIAL: NCT01333267
Title: Comparison of Skeletal and Mineral Metabolism Responses in Healthy African-Americans and Caucasians Using a Continuous Seven-Day Parathyroid Hormone (PTH) or Parathyroid Hormone-related Protein (PTHrP) Infusion
Brief Title: One Week Comparison Study of PTH and PTHrP Infusions
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Mara Horwitz, Associate Professor, University of Pittsburgh School of Medicine, University of Pittsburgh
Allocation: Non-Randomized | Model: Parallel | Masking: Single
Other Study IDs: PRO10060214
Record Dates: First submitted 2011-04-08; First posted 2011-04-11 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Osteoporosis; Hypercalcemia of Malignancy; Hyperparathyroidism; Bone Diseases, Endocrine
Keywords: Endocrine System Diseases; MusculoSkeletal System Disease; Hormones; Postmenopausal Women; Bone metabolism; Physiologic Properties; African-Americans
MeSH Terms: conditions — Osteoporosis; Humoral Hypercalcemia Of Malignancy; Hyperparathyroidism; Bone Diseases, Endocrine; Endocrine System Diseases; Musculoskeletal Diseases | interventions — parathyroid hormone-related peptide (1-36); Parathyroid Hormone; Parathyroid Hormone-Related Protein

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PTHrP group (Experimental): Subjects receive PTHrP(1-36) starting with doses of 2 picomoles (pmols)/kg/hr for one week. Subsequent dosing groups are determined by the response to PTHrP doses.
  Interventions: Drug: Parathyroid Hormone-related Protein (1-36); Drug: PTH (1-34) and PTHrP (1-36)
- PTH dosing group (Experimental): Subjects receive PTH(1-34) starting with doses of 2 picomoles (pmols)/kg/hr for one week. Subsequent dosing groups are determined by the response to PTH doses.
  Interventions: Drug: parathyroid hormone (1-34); Drug: PTH (1-34) and PTHrP (1-36)

INTERVENTIONS:
Drug: Parathyroid Hormone-related Protein (1-36) — PTHrP (1-36) intravenously at 2 picomoles (pmols)/kg/hr for one week; doses will be increased by 2 picomoles (pmols)/kg/hr in subsequent subjects.
  Other Names: PTHrP(1-36); Bone anabolic agents
  Arms: PTHrP group
Drug: parathyroid hormone (1-34) — PTH (1-34) intravenously at 2 picomoles (pmols)/kg/hr for one week; doses will be increased by 2 picomoles (pmols)/kg/hr in subsequent subjects.
  Other Names: PTH(1-34); Bone anabolic agent
  Arms: PTH dosing group
Drug: PTH (1-34) and PTHrP (1-36) — This is a dose escalation study to determine the maximum tolerable dose of Parathyroid Hormone-related Protein, PTHrP, or Parathyroid Hormone, PTH, that can be given safely over one week in healthy African-American volunteers. The investigators plan to infuse low doses of intravenous PTHrP or PTH to determine if it leads to a sustained and progressive suppression of bone formation as occurs in humoral hypercalcemia of malignancy (HHM) or an increase in bone formation as occurs in hyperparathyroidism (HPT). Additionally, the investigators will assess the direct influence of PTHrP and PTH on vitamin D metabolism, markers of bone turnover, and fractional excretion of calcium.
  Other Names: Parathyroid Hormone-related Protein (1-36); PTHrP(1-36); IND 49,175; Parathyroid Hormone (1-34); PTH (1-34); IND 60,979

SUMMARY:
This is a dose escalation study to determine the maximum tolerable dose of Parathyroid Hormone-related Protein, PTHrP, or Parathyroid Hormone, PTH, that can be given safely over one week in healthy African-American volunteers. The investigators plan to infuse low doses of intravenous PTHrP or PTH to determine if it leads to a sustained and progressive suppression of bone formation as occurs in humoral hypercalcemia of malignancy (HHM) or an increase in bone formation as occurs in hyperparathyroidism (HPT). Additionally, the investigators will assess the direct influence of PTHrP and PTH on vitamin D metabolism, markers of bone turnover, and fractional excretion of calcium. These results will be compared to previous studies of Caucasian volunteers.

DETAILED DESCRIPTION:
This study will expand upon earlier infusion studies in healthy Caucasian and Asian volunteers in which continuous infusions of PTH and PTHrP were given for six-, 12-, and 48 hours. These studies demonstrated: 1) There is a dose-related increase in 1,25 (OH)2 vitamin D in response to PTHrP and PTH over multiple days. 2) There is a markedly attenuated vitamin D response to PTHrP compared to PTH, particularly during the second 24 hours. 3) The increase in 1,25 (OH)2 vitamin D is almost certainly responsible for the greater calcemic effect of PTH compared to PTHrP. 4) PTHrP is obviously a weaker agonist of 1,25 (OH)2 vitamin D but does not result in its suppression as is seen in Humoral Hypercalcemia of Malignancy (HHM). Thus, the suppression of 1,25 (OH)2 vitamin D seen in HHM remains unexplained. In addition to assessing the effects of an infusion of PTHrP and PTH on calcium handling and 1,25 (OH)2 vitamin D, we also measured their effects on markers of bone turnover. Given the clinical observations seen in primary hyperparathyroidism (HPT) and HHM, we anticipated that PTH would stimulate both bone resorption and formation, while PTHrP would stimulate bone resorption but inhibit formation. However, we observed that infusions of PTHrP and PTH resulted in an equivalent, rapid increase in bone resorption as measured by N-telopeptide (NTx) and C-telopeptide (CTx), as well as a progressive decline in bone formation. There was no difference between PTH and PTHrP. Because of these findings, it was surmised that infusions of a longer duration would lead to an increase in bone formation and 1,25 (OH)2D production with both peptides, as is seen in HPT. Very recently, we have completed a seven-day infusion model in healthy Caucasian and Asian volunteers to test this hypothesis (J. Bone Min. Res., 2011). A total of 22 individuals were given either seven-day infusions of PTH or PTHrP, and maximal safe doses were found to be 2 and 4 picomoles (pmol)/kg/hour, respectively, lower than the doses used in previous, briefer infusion studies. All patients developed sustained but very mild hypercalcemia (mean = 10.3 mg/dL) and hypercalciuria with rapid increase in bone resorption. Surprisingly, bone formation again was suppressed for the entire seven days with a robust rebound in bone formation on cessation of the respective peptide. This is consistent with what may occur during lactation and HHM, but again contrary to what occurs in HPT.

The previous infusion studies were done only in Caucasian and Asian volunteers as there are extensively documented physiologic differences in bone metabolism between African-Americans and Caucasians. Much of the racial differences noted in bone metabolism come from the osteoporosis literature. African-Americans are known to have higher bone mineral densities (BMD) and to be at lower risk of developing fragility fractures. There are many factors which may explain these racial differences in bone metabolism, including altered calcium economy, vitamin D differences, peak attained bone mass, muscle mass and obesity, mechanism of falls, remodeling rates, bone micro-architecture, hip axis geometry, and other unknown hereditary differences. It is also well established that African-Americans on average, have lower 25-OH vitamin D concentrations and thus higher PTH levels. Despite elevations in PTH, there is paradoxically no increase in bone loss indicating that a relative skeletal resistance to PTH may exist. We hope that by performing this seven-day infusion protocol in healthy African-American volunteers we can learn more about racial differences in bone turnover, renal calcium, PTH concentrations, vitamin D metabolism, and skeletal responses to lactation in this under-studied population.

Ninety healthy African-American men and women will be screened for an eight-day inpatient admission to the Clinical & Translational Research Center (CTRC). Sixty evaluable research participants will receive a seven day infusion of a predetermined dose of either PTHrP or PTH. Vital signs and blood and urine tests will be monitored frequently as per the study flow sheet. The starting dose of either peptide, 2 picomoles (pmols)/kg, will be given to three normal healthy subjects. Via a dose escalation protocol, the dose will be escalated in increments with successive groups of three subjects each, until early adverse effects (mild hypercalcemia, postural hypotension, tachycardia) are seen. This determined safe dose will then be given to 10 subjects. This dose escalation study design has been used in several prior studies at this institution in order to achieve a sustained mild serum hypercalcemia in the 10.5-11 mg/dL range in research studies. The investigators with this study are trying to determine a safe dose of PTHrP and PTH in African-American volunteers and determining if this population has the same physiologic response as Caucasians.

Subject population will consist of healthy young African-American adults, ages 24-35. It is anticipated that we will need to screen 90 patients in order to obtain 60 evaluable subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy African-American subjects of both sexes between the ages of 24-35 years, who are able to spend one week on the Clinical & Translational Research Center (CTRC) at the University of Pittsburgh Medical Center (UPMC) Montefiore.

Exclusion Criteria:

* Subjects with cardiac, vascular, renal (serum creatinine > 1.5), pulmonary, endocrine, musculoskeletal, hepatic, hematologic, malignant, or rheumatologic disease will be excluded.
* Those found to have vitamin D deficiency, defined as a 25-OH vitamin D level < 10 ng/mL will also be excluded.
* Additionally, those with BMI > 30, anemia (hematocrit < 36% in women, <40% in men), significant alcohol use, illicit drug use, hypertension (BP>160/90), or baseline hypotension (systolic blood pressure < 90mmHg) will be excluded.
* Those taking chronic medications (except oral contraceptive pills (OCP's) or stable doses of thyroid replacement) or those who have received an investigational drug in the past 90 days will also be excluded.
* Prior participants in PTH or PTHrP studies will not be eligible to participate.
* Additionally pregnant women and lactating women will be excluded; all women will have a urine pregnancy test performed immediately before starting the study.

Ages: 24 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Safety: The absence of any dose limiting toxicity (DLT) criteria consisting of one major criteria or two minor criteria. | one week

SECONDARY OUTCOMES:
Blood collections analyzed for measurements of PTH(1-34), PTH(1-84), 25-OH vitamin D, 1,25(OH)2 vitamin D, markers of bone metabolism, and fractional excretion of calcium measurements. | one week

CONTACTS AND LOCATIONS:
Overall Officials: Mara J. Horwitz, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Dean T, Vilardaga JP, Potts JT Jr, Gardella TJ. Altered selectivity of parathyroid hormone (PTH) and PTH-related protein (PTHrP) for distinct conformations of the PTH/PTHrP receptor. Mol Endocrinol. 2008 Jan;22(1):156-66. doi: 10.1210/me.2007-0274. Epub 2007 Sep 13. PMID 17872377
- [Background] Horwitz MJ, Tedesco MB, Sereika SM, Syed MA, Garcia-Ocana A, Bisello A, Hollis BW, Rosen CJ, Wysolmerski JJ, Dann P, Gundberg C, Stewart AF. Continuous PTH and PTHrP infusion causes suppression of bone formation and discordant effects on 1,25(OH)2 vitamin D. J Bone Miner Res. 2005 Oct;20(10):1792-803. doi: 10.1359/JBMR.050602. Epub 2005 Jun 6. PMID 16160737
- [Background] Horwitz MJ, Tedesco MB, Sereika SM, Hollis BW, Garcia-Ocana A, Stewart AF. Direct comparison of sustained infusion of human parathyroid hormone-related protein-(1-36) [hPTHrP-(1-36)] versus hPTH-(1-34) on serum calcium, plasma 1,25-dihydroxyvitamin D concentrations, and fractional calcium excretion in healthy human volunteers. J Clin Endocrinol Metab. 2003 Apr;88(4):1603-9. doi: 10.1210/jc.2002-020773. PMID 12679445
- [Background] Nelson DA, Jacobsen G, Barondess DA, Parfitt AM. Ethnic differences in regional bone density, hip axis length, and lifestyle variables among healthy black and white men. J Bone Miner Res. 1995 May;10(5):782-7. doi: 10.1002/jbmr.5650100515. PMID 7639113
- [Background] George A, Tracy JK, Meyer WA, Flores RH, Wilson PD, Hochberg MC. Racial differences in bone mineral density in older men. J Bone Miner Res. 2003 Dec;18(12):2238-44. doi: 10.1359/jbmr.2003.18.12.2238. PMID 14672360
- [Background] Kalkwarf HJ, Zemel BS, Gilsanz V, Lappe JM, Horlick M, Oberfield S, Mahboubi S, Fan B, Frederick MM, Winer K, Shepherd JA. The bone mineral density in childhood study: bone mineral content and density according to age, sex, and race. J Clin Endocrinol Metab. 2007 Jun;92(6):2087-99. doi: 10.1210/jc.2006-2553. Epub 2007 Feb 20. PMID 17311856
- [Background] Hui SL, Dimeglio LA, Longcope C, Peacock M, McClintock R, Perkins AJ, Johnston CC Jr. Difference in bone mass between black and white American children: attributable to body build, sex hormone levels, or bone turnover? J Clin Endocrinol Metab. 2003 Feb;88(2):642-9. doi: 10.1210/jc.2002-020653. PMID 12574194
- [Background] Bachrach LK, Hastie T, Wang MC, Narasimhan B, Marcus R. Bone mineral acquisition in healthy Asian, Hispanic, black, and Caucasian youth: a longitudinal study. J Clin Endocrinol Metab. 1999 Dec;84(12):4702-12. doi: 10.1210/jcem.84.12.6182. PMID 10599739
- [Background] Gilsanz V, Skaggs DL, Kovanlikaya A, Sayre J, Loro ML, Kaufman F, Korenman SG. Differential effect of race on the axial and appendicular skeletons of children. J Clin Endocrinol Metab. 1998 May;83(5):1420-7. doi: 10.1210/jcem.83.5.4765. PMID 9589632
- [Background] Abrams SA, O'brien KO, Liang LK, Stuff JE. Differences in calcium absorption and kinetics between black and white girls aged 5-16 years. J Bone Miner Res. 1995 May;10(5):829-33. doi: 10.1002/jbmr.5650100521. PMID 7639119
- [Background] Gilsanz V, Roe TF, Mora S, Costin G, Goodman WG. Changes in vertebral bone density in black girls and white girls during childhood and puberty. N Engl J Med. 1991 Dec 5;325(23):1597-600. doi: 10.1056/NEJM199112053252302. PMID 1944449
- [Background] Luckey MM, Wallenstein S, Lapinski R, Meier DE. A prospective study of bone loss in African-American and white women--a clinical research center study. J Clin Endocrinol Metab. 1996 Aug;81(8):2948-56. doi: 10.1210/jcem.81.8.8768857.
- [Background] Thomas PA. Racial and ethnic differences in osteoporosis. J Am Acad Orthop Surg. 2007;15 Suppl 1:S26-30. doi: 10.5435/00124635-200700001-00008. PMID 17766786
- [Background] Han ZH, Palnitkar S, Rao DS, Nelson D, Parfitt AM. Effects of ethnicity and age or menopause on the remodeling and turnover of iliac bone: implications for mechanisms of bone loss. J Bone Miner Res. 1997 Apr;12(4):498-508. doi: 10.1359/jbmr.1997.12.4.498. PMID 9101361
- [Background] Cauley JA, Wampler NS, Barnhart JM, Wu L, Allison M, Chen Z, Hendrix S, Robbins J, Jackson RD; Women's Health Initiative Observational Study. Incidence of fractures compared to cardiovascular disease and breast cancer: the Women's Health Initiative Observational Study. Osteoporos Int. 2008 Dec;19(12):1717-23. doi: 10.1007/s00198-008-0634-y. Epub 2008 Jul 16. PMID 18629572
- [Background] Cauley JA, Palermo L, Vogt M, Ensrud KE, Ewing S, Hochberg M, Nevitt MC, Black DM. Prevalent vertebral fractures in black women and white women. J Bone Miner Res. 2008 Sep;23(9):1458-67. doi: 10.1359/jbmr.080411. PMID 18442309
- [Background] Cauley JA, Lui LY, Ensrud KE, Zmuda JM, Stone KL, Hochberg MC, Cummings SR. Bone mineral density and the risk of incident nonspinal fractures in black and white women. JAMA. 2005 May 4;293(17):2102-8. doi: 10.1001/jama.293.17.2102. PMID 15870413
- [Background] Opotowsky AR, Bilezikian JP. Racial differences in the effect of early milk consumption on peak and postmenopausal bone mineral density. J Bone Miner Res. 2003 Nov;18(11):1978-88. doi: 10.1359/jbmr.2003.18.11.1978. PMID 14606510
- [Background] Cosman F, Nieves J, Dempster D, Lindsay R. Vitamin D economy in blacks. J Bone Miner Res. 2007 Dec;22 Suppl 2:V34-8. doi: 10.1359/jbmr.07s220. PMID 18290719
- [Background] Harris SS, Soteriades E, Dawson-Hughes B; Framingham Heart Study; Boston Low-Income Elderly Osteoporosis Study. Secondary hyperparathyroidism and bone turnover in elderly blacks and whites. J Clin Endocrinol Metab. 2001 Aug;86(8):3801-4. doi: 10.1210/jcem.86.8.7783. PMID 11502814
- [Background] Cosman F, Morgan DC, Nieves JW, Shen V, Luckey MM, Dempster DW, Lindsay R, Parisien M. Resistance to bone resorbing effects of PTH in black women. J Bone Miner Res. 1997 Jun;12(6):958-66. doi: 10.1359/jbmr.1997.12.6.958. PMID 9169356
- [Background] Fuleihan GE, Gundberg CM, Gleason R, Brown EM, Stromski ME, Grant FD, Conlin PR. Racial differences in parathyroid hormone dynamics. J Clin Endocrinol Metab. 1994 Dec;79(6):1642-7. doi: 10.1210/jcem.79.6.7989469.
- [Background] Aloia JF, Patel M, Dimaano R, Li-Ng M, Talwar SA, Mikhail M, Pollack S, Yeh JK. Vitamin D intake to attain a desired serum 25-hydroxyvitamin D concentration. Am J Clin Nutr. 2008 Jun;87(6):1952-8. doi: 10.1093/ajcn/87.6.1952. PMID 18541590
- [Background] Aloia JF. African Americans, 25-hydroxyvitamin D, and osteoporosis: a paradox. Am J Clin Nutr. 2008 Aug;88(2):545S-550S. doi: 10.1093/ajcn/88.2.545S. PMID 18689399
- [Background] Aloia JF, Talwar SA, Pollack S, Feuerman M, Yeh JK. Optimal vitamin D status and serum parathyroid hormone concentrations in African American women. Am J Clin Nutr. 2006 Sep;84(3):602-9. doi: 10.1093/ajcn/84.3.602. PMID 16960175
- [Background] Aloia JF, Talwar SA, Pollack S, Yeh J. A randomized controlled trial of vitamin D3 supplementation in African American women. Arch Intern Med. 2005 Jul 25;165(14):1618-23. doi: 10.1001/archinte.165.14.1618. PMID 16043680
- [Background] Barrett-Connor E, Siris ES, Wehren LE, Miller PD, Abbott TA, Berger ML, Santora AC, Sherwood LM. Osteoporosis and fracture risk in women of different ethnic groups. J Bone Miner Res. 2005 Feb;20(2):185-94. doi: 10.1359/JBMR.041007. Epub 2004 Oct 18. PMID 15647811
- [Background] Cauley JA, Wu L, Wampler NS, Barnhart JM, Allison M, Chen Z, Jackson R, Robbins J. Clinical risk factors for fractures in multi-ethnic women: the Women's Health Initiative. J Bone Miner Res. 2007 Nov;22(11):1816-26. doi: 10.1359/jbmr.070713. PMID 17638574
- [Background] Faulkner KA, Cauley JA, Zmuda JM, Landsittel DP, Nevitt MC, Newman AB, Studenski SA, Redfern MS. Ethnic differences in the frequency and circumstances of falling in older community-dwelling women. J Am Geriatr Soc. 2005 Oct;53(10):1774-9. doi: 10.1111/j.1532-5415.2005.53514.x. PMID 16181179
- [Background] Finkelstein JS, Lee ML, Sowers M, Ettinger B, Neer RM, Kelsey JL, Cauley JA, Huang MH, Greendale GA. Ethnic variation in bone density in premenopausal and early perimenopausal women: effects of anthropometric and lifestyle factors. J Clin Endocrinol Metab. 2002 Jul;87(7):3057-67. doi: 10.1210/jcem.87.7.8654. PMID 12107201
- [Background] Schnitzler CM, Mesquita JM. Cortical bone histomorphometry of the iliac crest in normal black and white South African adults. Calcif Tissue Int. 2006 Dec;79(6):373-82. doi: 10.1007/s00223-006-0053-z. Epub 2006 Dec 8. PMID 17160576
- [Background] Cummings SR, Cauley JA, Palermo L, Ross PD, Wasnich RD, Black D, Faulkner KG. Racial differences in hip axis lengths might explain racial differences in rates of hip fracture. Study of Osteoporotic Fractures Research Group. Osteoporos Int. 1994 Jul;4(4):226-9. doi: 10.1007/BF01623243. PMID 7949753
- [Background] Perry HM 3rd, Horowitz M, Morley JE, Fleming S, Jensen J, Caccione P, Miller DK, Kaiser FE, Sundarum M. Aging and bone metabolism in African American and Caucasian women. J Clin Endocrinol Metab. 1996 Mar;81(3):1108-17. doi: 10.1210/jcem.81.3.8772584.
- [Background] Jacobsen SJ, Goldberg J, Miles TP, Brody JA, Stiers W, Rimm AA. Race and sex differences in mortality following fracture of the hip. Am J Public Health. 1992 Aug;82(8):1147-50. doi: 10.2105/ajph.82.8.1147. PMID 1636840
- [Background] Mikuls TR, Saag KG, George V, Mudano AS, Banerjee S. Racial disparities in the receipt of osteoporosis related healthcare among community-dwelling older women with arthritis and previous fracture. J Rheumatol. 2005 May;32(5):870-5. PMID 15868624
- [Background] Alam NM, Archer JA, Lee E. Osteoporotic fragility fractures in African Americans: under-recognized and undertreated. J Natl Med Assoc. 2004 Dec;96(12):1640-5. PMID 15624249
- [Background] Looker AC. The skeleton, race, and ethnicity. J Clin Endocrinol Metab. 2002 Jul;87(7):3047-50. doi: 10.1210/jcem.87.7.8779. No abstract available. PMID 12107199
- [Background] Bell NH, Bilezikian JP, Bone HG 3rd, Kaur A, Maragoto A, Santora AC; MK-063 Study Group. Alendronate increases bone mass and reduces bone markers in postmenopausal African-American women. J Clin Endocrinol Metab. 2002 Jun;87(6):2792-7. doi: 10.1210/jcem.87.6.8575. PMID 12050252
- [Background] Neer RM, Arnaud CD, Zanchetta JR, Prince R, Gaich GA, Reginster JY, Hodsman AB, Eriksen EF, Ish-Shalom S, Genant HK, Wang O, Mitlak BH. Effect of parathyroid hormone (1-34) on fractures and bone mineral density in postmenopausal women with osteoporosis. N Engl J Med. 2001 May 10;344(19):1434-41. doi: 10.1056/NEJM200105103441904. PMID 11346808
- [Background] Lau EM, Suriwongpaisal P, Lee JK, Das De S, Festin MR, Saw SM, Khir A, Torralba T, Sham A, Sambrook P. Risk factors for hip fracture in Asian men and women: the Asian osteoporosis study. J Bone Miner Res. 2001 Mar;16(3):572-80. doi: 10.1359/jbmr.2001.16.3.572. PMID 11277276
- [Background] Awumey EM, Mitra DA, Hollis BW, Kumar R, Bell NH. Vitamin D metabolism is altered in Asian Indians in the southern United States: a clinical research center study. J Clin Endocrinol Metab. 1998 Jan;83(1):169-73. doi: 10.1210/jcem.83.1.4514. PMID 9435436
- [Background] Looker AC, Orwoll ES, Johnston CC Jr, Lindsay RL, Wahner HW, Dunn WL, Calvo MS, Harris TB, Heyse SP. Prevalence of low femoral bone density in older U.S. adults from NHANES III. J Bone Miner Res. 1997 Nov;12(11):1761-8. doi: 10.1359/jbmr.1997.12.11.1761. PMID 9383679
- [Background] Wright NM, Papadea N, Willi S, Veldhuis JD, Pandey JP, Key LL, Bell NH. Demonstration of a lack of racial difference in secretion of growth hormone despite a racial difference in bone mineral density in premenopausal women--a Clinical Research Center study. J Clin Endocrinol Metab. 1996 Mar;81(3):1023-6. doi: 10.1210/jcem.81.3.8772569.
- [Background] Heaney RP. Bone mass, the mechanostat, and ethnic differences. J Clin Endocrinol Metab. 1995 Aug;80(8):2289-90. doi: 10.1210/jcem.80.8.7629221. No abstract available.
- [Background] Cundy T, Cornish J, Evans MC, Gamble G, Stapleton J, Reid IR. Sources of interracial variation in bone mineral density. J Bone Miner Res. 1995 Mar;10(3):368-73. doi: 10.1002/jbmr.5650100306. PMID 7785457
- [Background] Wright NM, Renault J, Willi S, Veldhuis JD, Pandey JP, Gordon L, Key LL, Bell NH. Greater secretion of growth hormone in black than in white men: possible factor in greater bone mineral density--a clinical research center study. J Clin Endocrinol Metab. 1995 Aug;80(8):2291-7. doi: 10.1210/jcem.80.8.7543111.
- [Background] Looker AC, Johnston CC Jr, Wahner HW, Dunn WL, Calvo MS, Harris TB, Heyse SP, Lindsay RL. Prevalence of low femoral bone density in older U.S. women from NHANES III. J Bone Miner Res. 1995 May;10(5):796-802. doi: 10.1002/jbmr.5650100517. PMID 7639115
- [Background] Looker AC, Wahner HW, Dunn WL, Calvo MS, Harris TB, Heyse SP, Johnston CC Jr, Lindsay RL. Proximal femur bone mineral levels of US adults. Osteoporos Int. 1995;5(5):389-409. doi: 10.1007/BF01622262. PMID 8800790
- [Background] Villa ML. Cultural determinants of skeletal health: the need to consider both race and ethnicity in bone research. J Bone Miner Res. 1994 Sep;9(9):1329-32. doi: 10.1002/jbmr.5650090902. No abstract available. PMID 7817815
- [Background] Baron JA, Barrett J, Malenka D, Fisher E, Kniffin W, Bubolz T, Tosteson T. Racial differences in fracture risk. Epidemiology. 1994 Jan;5(1):42-7. doi: 10.1097/00001648-199401000-00008. PMID 8117781
- [Background] Silverman SL, Madison RE. Decreased incidence of hip fracture in Hispanics, Asians, and blacks: California Hospital Discharge Data. Am J Public Health. 1988 Nov;78(11):1482-3. doi: 10.2105/ajph.78.11.1482. PMID 3177728
- [Background] Looker AC, Flegal KM, Melton LJ 3rd. Impact of increased overweight on the projected prevalence of osteoporosis in older women. Osteoporos Int. 2007 Mar;18(3):307-13. doi: 10.1007/s00198-006-0241-8. Epub 2006 Oct 20. PMID 17053871